CLINICAL TRIAL: NCT06428266
Title: Comparative Study of Safety and Efficacy of Closed Dacryointubation vs Bicanalicular Intubation in the Treatment of Proximal Tear Duct Obstruction in Adult Patients
Brief Title: Closed Dacryointubation vs Bicanalicular Intubation for Proximal Tear Duct Obstruction
Acronym: DICvsBIcanal
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto de Oftalmología Fundación Conde de Valenciana (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CI 09 015 008
Record Dates: First submitted 2024-05-20; First posted 2024-05-24 (Actual); Last update posted 2024-05-31 (Actual); Status verified 2024-05

CONDITIONS: Lacrimal Duct Obstruction; Lacrimal Apparatus Diseases; Lacrimal Stenosis; Lacrimal Elimination
Keywords: upper lacrimal duct obstruction; bicanalicular intubation; closed dacriointubation
MeSH Terms: conditions — Lacrimal Duct Obstruction; Lacrimal Apparatus Diseases

STUDY DESIGN:
Intervention Model Description: Patients from the consultation of the Oculoplastics Department of the Institute of Ophthalmology "Conde de Valenciana I.A.P", between July 2021 and July 2022 who met the inclusion and exclusion criteria were enrolled
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Closed dacryointubation (Active Comparator): Patients undergoing conventional closed dacryointubation with Crawford's tube
  Interventions: Procedure: Closed dacryointubation
- Bicanalicular Intubation (Experimental): Patients undergoing bicanalicular intubation with Self-Stable Intubation Set II FCI
  Interventions: Device: Bicanalicular intubation

INTERVENTIONS:
Device: Bicanalicular intubation — Placement of the bicanalicular intubation set at each lacrimal point and fixed by means of its flaps at the level of the opening of the lacrimal sac.
  Arms: Bicanalicular Intubation
Procedure: Closed dacryointubation — Placement of dacryointubation tube through the canaliculus until it reaches the medial wall of the lacrimal sac and then passed the nasolacrimal duct until it empties out at the level of the inferior meatus.
  Arms: Closed dacryointubation

SUMMARY:
In Mexico, upper lacrimal duct obstruction (ULDO) is a common pathology, and the standard surgical treatment is closed dracryointubation. Based on statistics from our headquarters, in 30% of cases there is a failure of the technique and recurrence of symptoms due to associated complications. Because of this, the application of a self-stable bicananlicular intubation set is proposed. The aim of this study is to describe the difference in efficacy and complication rate between the application of the self-stable bicanalicular intubation set II (FCI) and closed dacryointubation in patients with ULDO .

DETAILED DESCRIPTION:
Upper lacrimal duct obstruction (ULDO) or proximal lacrimal tract obstruction occurs when an occlusion is located in the lacrimal point, in superior and inferior canaliculi, or in the common canaliculus. When the ULDO is at the level of the canaliculi (superior, inferior or common), the alternatives available for its management are closed dacryointubation with Crowford catheter, conjunctivadacryocystorhinostomy, and bicanalicular intubation.

Closed dacryointubation with Crowford tube is a technique effective in approximately 90% of children diagnosed with congenital occlusion of the lacrimal duct, however, in adults the reported surgical success rate is lower, approximately 70% according to different authors.

The conjunctivadacryocystorhinostomy is the procedure proposed by many authors when there is point and canaliculi obstruction in which canalicular intubation cannot be performed due to atresia or total obstruction.

The bicanaliculalr intubation with the Self-Stable Canalicular Intubation Set (FCI R), an FDA-approved silicone bicanalicular retention device, is especially indicated for the treatment of lacrimal point stenosis and horizontal canalicular obstruction.

The aim of this study is to describe the difference in efficacy and complication rate between the application of the self-stable bicanalicular intubation set II (ICF) and closed dacryointubation in patients with ULDO

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years of age
* Patients with stenosis and incomplete obstruction of the upper lacrimal duct with epiphora > 2 on the Munk scale who have not previously undergone surgery on the affected tear duct
* Patients who may undergo general anesthesia and sedation
* Patients who are able to present and continue follow-up for the duration of the study
* Acceptance to participate in the study by signing an informed consent

Exclusion Criteria:

* Patients with ocular surface involvement affecting the upper lacrimal duct, such as blepharitis with tear point epithelialization
* Patients with lacrimal point malposition and/or eyelid malposition due to entropion or ectropion
* Patients with congenital or acquired obstruction of the lower lacrimal duct
* Patients with a history of facial paralysis
* Patients with systemic inflammatory disease such as scarring pemphigoid or Steven Johnson
* Patients in whom tumour involvement of the lacrimal duct is suspected
* Patients with reflex tear hypersecretion due to ocular surface involvement or other causes.
* Pregnancy and breastfeeding
* Active infection, eye trauma, history of facial trauma with broken bones of the nose, or history of sinus surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-07-31 (Actual)

PRIMARY OUTCOMES:
Irrigation of tha lacrimal duct | three and four months after the procedure
  Irrigation of the lacrimal duct with saline solution to seek for permeability
Epiphora | one, three and four months after surgery
  evidence of epiphora as told by the subject

SECONDARY OUTCOMES:
Occurrence of epistaxis | one, three and four months after surgery
  postoperative bleeding throug the nose
Presence of extrusion of bicanalicular intubation tubes | one, three and four months after surgery
  extruded or non-extruded
How well is the positioning of the silicone tubes | one, three and four months after surgery
  how well positioned or poorly positioned the tubes are

CONTACTS AND LOCATIONS:
Locations (1):
- Institiuto de Oftalmología Fundación Conde de Valenciana, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] 1. Schaefer DP. Acquired Etiologies of Lacrimal System Obstructions. In: Cohen AJ, Mercandetti M, Brazzo BG, editors. The Lacrimal System [Internet]. Springer New York; 2006 [cited 2020 Jan 15]. p. 43-65.
- [Background] Fulcher T, O'Connor M, Moriarty P. Nasolacrimal intubation in adults. Br J Ophthalmol. 1998 Sep;82(9):1039-41. doi: 10.1136/bjo.82.9.1039. PMID 9893595
- [Background] Pashby RC, Rathbun JE. Silicone tube intubation of the lacrimal drainage system. Arch Ophthalmol. 1979 Jul;97(7):1318-22. doi: 10.1001/archopht.1979.01020020060014. PMID 454271
- [Background] Tabatabaie SZ, Rajabi MT, Rajabi MB, Eshraghi B. Randomized study comparing the efficacy of a self-retaining bicanaliculus intubation stent with Crawford intubation in patients with canalicular obstruction. Clin Ophthalmol. 2012;6:5-8. doi: 10.2147/OPTH.S25172. Epub 2011 Dec 20. PMID 22259230
- See also: characteristics of the Self-Stable Intubation Set II FCI — http://www.accessdata.fda.gov/cdrh_docs/pdf13/K130375.pdf